CLINICAL TRIAL: NCT06493435
Title: Evaluation du Protocole de PBM du Service de Chirurgie gynécologique du CHU d'Angers: étude Periope 2
Brief Title: Efficiency of Patient Blood Management Protocol in Gynecological Surgery Department (PERIOPESGYNECO)
Acronym: PERIOPESGYNECO
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 24_0207
Record Dates: First submitted 2024-06-18; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-06

CONDITIONS: Anemia
Keywords: anemia; perioperative period; post operative recovery; patient blood management
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Perioperative anemia is associated with higher risk of red blood cell transfusion, higher rates of morbimortality and lower quality of postoperative recovery. In a context of focussing on higher quality management and improved recovery after surgery, development of Patient Blood management has increased. This study aim to assess PBM protocole in a postoperative context of gynaecological surgery, by comparing indicators at two time periods: 2 and 8 months after establishment of PBM protocol.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* being hospitalised for planned hysterectomy or cancer related ovariectomy

Exclusion Criteria:

* less than 18 years
* non french speaker
* being under a legal individual protection measure
* not being able to consent
* being opposed to data collection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with planned surgery of hyterectomy or cancer related ovariectomy
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of immediate pre operative anemia | at 2 and 8 months after establishment of PBM protocol
  preoperative Hb<13g/dL

SECONDARY OUTCOMES:
rate of preoperative anemia that need to be treated diagnosed during anesthetic consultation | at 2 and 8 months after establishment of PBM protocol
  Hb<13 g/dL
rate of Hemoglobin dosage available during anesthetic evaluation | at 2 and 8 months after establishment of PBM protocol
  number and rate of blood analyses
rate of preoperative iron deficiency that need to be treated diagnosed during anesthetic consultation | at 2 and 8 months after establishment of PBM protocol
  blood ferritin level <100 ng/mL
adequacy between diagnosed iron deficiency anemia and treatment | at 2 and 8 months after establishment of PBM protocol
  rate of iron prescription
effectiveness of iron treatment | at 2 and 8 months after establishment of PBM protocol
  rate of persistent pre operative anemia after iron treatment
immediat effect of surgery on anemia incidence | at 2 and 8 months after establishment of PBM protocol
  rate of post operative anemia (Hb<12g/dL)/ rate of post operative iron treatment
delayed effect of surgery on anemia incidence | at 2 and 8 months after establishment of PBM protocol
  rate of delayed post operative anemia or iron deficiency
early post operative recovery | at 2 and 8 months after establishment of PBM protocol
  FQoR 15 on the day of hospital dischage
delayed post operative recovery | at 2 and 8 months after establishment of PBM protocol
  FQoR 15 at the post operative surgical visit
adhesion to PBM protocol (rate of anemia) | at 2 and 8 months after establishment of PBM protocol
  comparison of rate of anemia screening
efficiency of PBM protocol (iron treatment rate) | at 2 and 8 months after establishment of PBM protocol
  comparison of iron treatment rate
adhesion to PBM protocol (missing datas) | at 2 and 8 months after establishment of PBM protocol
  comparison of the rate of missing datas
efficiency of PBM protocol (preoperative anemia rate) | at 2 and 8 months after establishment of PBM protocol
  comparison of the rate of preoperative anemia
efficiency of PBM protocol (perioperative transfusion rate) | at 2 and 8 months after establishment of PBM protocol
  comparison of the rate of peri opeartive transfusion
efficiency of PBM protocol (mean of FQoR-15) | at 2 and 8 months after establishment of PBM protocol
  comparison of the mean of FQoR-15
efficiency of PBM protocol (mean of FQoR-15 between patients with or without preoperative anemia) | at 2 and 8 months after establishment of PBM protocol
  comparison of FQoR-15 means between patients with or without preoperative anemia
efficiency of PBM protocol (rate of screening anemia and the rate of preoperative anemia ) | at 2 and 8 months after establishment of PBM protocol
  comparison of the rate of screening anemia and the rate of preoperative anemia
efficiency of PBM protocol (Hb level between anesthetic evaluation and pre anesthetic visit) | at 2 and 8 months after establishment of PBM protocol
  comparison of Hb level between anesthetic evaluation and pre anesthetic visit (paired T test)
efficiency of PBM protocol (difference of hemoglobin level after iron treatment) | at 2 and 8 months after establishment of PBM protocol
  mean difference of hemoglobin level after iron treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sigismond Lasocki, Principal Investigator — University Hospital, Angers

IPD SHARING:
Plan to Share IPD: No